CLINICAL TRIAL: NCT01609959
Title: Effects of the New Angiotensin II Receptor Blocker Azilsartan Versus Valsartan on Blood Pressure in Japanese Patients With Hypertension
Brief Title: New Angiotensin II Receptor Blocker Azilsartan Study for Stronger Blood Pressure Lowering
Acronym: NARA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nara Medical University (Other)
Responsible Party: Principal Investigator, Yoshihiko Saito, Professor, Nara Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-Ken-001
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Hypertension
Keywords: Hypertension; Angiotensin II Receptor Blocker; Azilsartan; Valsartan
MeSH Terms: conditions — Hypertension | interventions — azilsartan; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azilsartan group (Active Comparator)
  Interventions: Drug: Azilsartan
- Valsartan group (Active Comparator)
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Azilsartan — Azilsartan 20 mg or 40 mg (if blood pressure does not reach the target after 6 weeks) per day for 12 weeks
  Arms: Azilsartan group
Drug: Valsartan — Valsartan 160 mg per day
  Arms: Valsartan group

SUMMARY:
The purpose of this study is to compare blood pressure lowering effect of azilsartan with that of valsartan in Japanese patients with hypertension who have already taken normal-dose angiotensin II receptor blockers.

DETAILED DESCRIPTION:
Hypertension plays a major role in the development of cardiovascular disease. Several guidelines require strict control of blood pressure for preventing cardiovascular events; however, the control is often poor.

A new angiotensin II receptor blocker (ARB), azilsartan, is the first drug which is superior to other ARBs in blood pressure lowering in phase III clinical trials in Japan. We try to evaluate effect of azilsartan on blood pressure lowering in Japanese patients with hypertension who have already taken normal-dose ARBs, and to compare it with that of valsartan.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients treated with normal-dose angiotensin II receptor blockers (ARBs) in Japan
* Normal-dose ARBs in Japan are defined as follows: losartan potassium 50 mg, candesartan cilexetil 8 mg, valsartan 80 mg, telmisartan 40 mg, olmesartan medoxomil 20 mg, or irbesartan 100mg per day.

Exclusion Criteria:

* Hypersensitivity for azilsartan and valsartan
* Pregnant female
* History of azilsartan use within 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in Office Blood Pressure | Baseline and every 2 weeks (up to 12 weeks)
  Change in blood pressure measured at a clinic

SECONDARY OUTCOMES:
Change in Home Blood Pressure | Baseline and every 2 weeks (up to 12 weeks)
  Change in blood pressure measured at home
  Blood pressure is measured twice daily in the morning fasting before taking any drugs.
Change in Renal Function | Baseline and 12 weeks
  Changes in levels of serum creatinine and proteinuria
Change in Fasting Triglyceride | Baseline and 12 weeks
Change in Glycemic Control | Baseline and 12 weeks
  Changes in levels of fasting blood glucose, hemogrobin A1C and fasting insulin (if needed)
Change in Plasma Aldosterone Concentration | Baseline and 12 weeks
  Only in patients with secondary hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihiko Saito, MD, PhD, Principal Investigator — First Department of Internal Medicine, Nara Medical University
Locations (1):
- First Department of Nara Medical University, Kashihara, Nara, Japan